CLINICAL TRIAL: NCT00558870
Title: Role of Methadone As Co-Opioid Analgesic in Cancer Patients
Brief Title: Role of Methadone As Co-Opioid Analgesic
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006-0641; NCI-2012-01553 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-11-14; First posted 2007-11-15 (Estimated); Results first posted 2016-04-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Pain
Keywords: Solid Tumors; Morphine; Methadone; Co-Opioid Analgesic; Pain
MeSH Terms: conditions — Pain | interventions — Morphine; Methadone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Morphine Only (Active Comparator): Morphine - Arm 1: 2 Doses of "Slow-Release" Morphine PO Every 12 Hours, Every Day for 15 Days (plus or minus 3 days)."Immediate-release" morphine may be used, if needed, for pain.
  Interventions: Drug: Morphine
- Morphine + Methadone (Active Comparator): Arm 2: 1 Dose of Slow-Release Morphine PO Every 12 Hours, Every Day for 15 Days (plus or minus 3 days).)."Immediate-release" morphine may be used, if needed, for pain.
  1 Dose of Methadone PO Every 12 Hours, Every Day for 15 Days (plus or minus 3 days)
  Interventions: Drug: Morphine; Drug: Methadone

INTERVENTIONS:
Drug: Morphine — Arm 1: 2 Doses of "Slow-Release" Morphine PO Every 12 Hours, Every Day for 15 Days (plus or minus 3 days)."Immediate-release" morphine may be used, if needed, for pain.
Drug: Methadone — 1 Dose of Methadone PO Every 12 Hours, Every Day for 15 Days (plus or minus 3 days)
  Arm 2: 1 Dose of Slow-Release Morphine PO Every 12 Hours, Every Day for 15 Days (plus or minus 3 days).)."Immediate-release" morphine may be used, if needed, for pain.
  Arms: Morphine + Methadone

SUMMARY:
Objectives:

Primary Objective:

To determine whether the addition of low dose methadone to morphine(in the methadone group) has a lower dose escalation index as compared to the morphine alone(in the morphine group) at Day 15 (+/- 3 days)

Secondary Objectives:

To determine whether individuals on the methadone arm have lower pain intensity than the morphine alone arm as demonstrated by a decrease in two points from baseline (+/- 3 days) in their ESAS score at Day 15 (+/- 3 days).

To determine whether the methadone group of experiences fewer opioid induced neurotoxic side effects (including sedation, myoclonus, hallucinations, hyperalgesia and confusion) as compared to the morphine alone group at Day 15 (+/- 3 days).

DETAILED DESCRIPTION:
The Study Drugs:

Methadone and morphine are both designed to block pain receptors (cells that are sensitive to particular drugs) in your nerves and brain.

Study Groups and Study Drug Administration:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in toss of a coin) to 1 of 2 groups. Participants in Group 1 will stay on morphine only. Participants in Group 2 will receive morphine plus methadone. You will have an equal chance (50/50) of being placed in either of the 2 groups. You, the medical staff, and study researchers will not know which group you have been assigned to. If necessary, your doctor will be able to find out what group you are in the event of an emergency.

Participants in Group 1 will take 2 doses of "slow-release" morphine by mouth every 12 hours, every day for 15 days (plus or minus 3 days). You will also have access to "immediate-release" morphine to be used, as needed, for pain. If you need more than 3 of these immediate-release doses in a 24-hour period, you should call your study doctor.

Participants in Group 2 will take 1 dose of slow-release morphine and 1 dose of methadone by mouth every 12 hours, every day for 15 days (plus or minus 3 days). You will also have access to immediate-release morphine to be used, as needed, for pain. If you need more than 3 of these immediate-release doses in a 24-hour period, you should call your study doctor.

You will complete a questionnaire once daily about symptoms and pain you may be experiencing. It will take about 5 minutes to complete each time.

You will be provided with a drug diary to write down when and how often you take pain medication.

Study Visits:

On Days 8 and 15 (plus or minus 3 days) the following test and procedures will be performed:

* You will complete 3 questionnaires about any side effects you may be having. They will take about 15-20 minutes to complete.
* You will have tests to see how sensitive your skin is.

On Day 15 only (plus or minus 3 days), you will have blood (about 1 teaspoon) drawn to measure kidney function.

Length of Study:

You will be off-study after Day 15 (plus or minus 3 days). You will be taken off study early if the disease gets worse or intolerable side effects occur.

This is an investigational study. Methadone and morphine are both FDA approved and commercially available. Their use together is investigational. Up to 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Individual reporting average pain score for the last 24 hours that is at least a 4 on a numerical scale from 0 to 10 (0= no pain, 10=the worst possible pain) with a history of cancer (active or no evidence of disease).
2. Individual is receiving strong opioids (morphine, fentanyl, oxycodone, hydromorphone) for 3 weeks prior to enrollment.
3. Individual requires at least 150 mg of daily morphine equivalent daily dose for cancer pain. Using the formula MEDD = dose X MEDD Factor (App L) it would be follows: morphine: a 24 hour total oral intake (sum of PRN and around the clock doses) of 150 mg or greater would qualify the patient, for fentanyl alone: a 24 hour total transdermal intake of 75mcg/h or greater would qualify the patient, for oxycodone alone: a 24 hour total oral intake of 100 mg or greater would qualify the patient, and for hydromorphone alone: a 24 hour total oral intake of 30 mg/day or greater would qualify the patient.
4. Individual has the ability to receive morphine or methadone orally.
5. Individual has no known allergy of history of severe toxicity to morphine or methadone.
6. Individual has normal cognition defined as normal state of arousal and absence of obvious clinical findings of confusion, memory or concentration deficit.
7. Individual has adequate renal function (creatinine less or equal to 2.0 MG/DL)
8. Individual has a Zubrod performance status of 3 or lower.
9. Individual is willing to sign written informed consent.
10. Individual is 18 years of age or older.
11. Individual on stable doses(on same dose for at least one week) of nonopioid analgesics including NSAIDS, corticosteroids, gabapentin, pregabalin, or antidepressants prescribed for the purposes of pain control.

Exclusion Criteria:

1. Individual is determined incapable of completing the evaluation forms.
2. Individual with clinically evident impaired cognition.
3. Patient with MEDD greater than 600.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Yennurajalingam, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: November 13, 2007 to August 26, 2010. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Study was halted early due to slow accrual. One participant of the five enrolled did not get randomized therefore did not receive treatment and is excluded.
Groups:
- Morphine Only: 2 Doses oral Slow-Release Morphine (7.5 mg) every 12 hours for 15 Days, and immediate-release morphine, if needed, for breakthrough pain.
- Morphine + Methadone: 1 Dose oral Slow-Release Morphine (7.5 mg) plus oral Methadone dose (starting dose 2.5 mg) every 12 hours for 15 Days. Immediate-release morphine, if needed, for breakthrough pain.
Period: Overall Study
Arm/Group | Morphine Only | Morphine + Methadone
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morphine Only | Morphine + Methadone | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Median (Full Range); unit: years] | 45 [42 to 48] | 35 [28 to 42] | 42 [28 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response (OR)
Description: Objective response (OR) is defined as a dose escalation index <20 where Opioid escalation index measured in milligrams is calculated by the formula, (OMD-OSD)/days, OMD = Opioid maximum dose as expressed in equianalgesic dose of oral morphine in milligrams, OSD= Opioid starting dose at the time of referral to palliative care/ pain specialist for the treatment of cancer pain as expressed in equianalgesic dose of oral morphine in milligrams. A low index indicates the achievement of adequate analgesia or appearance of uncontrollable side effects limiting upward titration over time. OR used in determining whether the addition of low dose methadone to morphine (in the methadone group) has a lower dose escalation index as compared to the morphine alone (in the morphine group) at Day 15.
Time Frame: Day 15 (+/- 3 days)
Population: There were no participants analyzed in each group for outcome variable; the study was terminated without completing any analysis because the sample size was too small to detect any differences between the groups.
Arm/Group | Morphine Only | Morphine + Methadone
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Dose Escalation Index at Day 15 (+/- 3 Days)
Description: Intended index period from baseline to Day 15 to determine whether the addition of low dose methadone to morphine (in the methadone group) has a lower dose escalation index as compared to the morphine alone (in the morphine group) at Day 15 (+/- 3 days). To determine whether the methadone group of individuals has a lower dose escalation index as compared to the morphine alone group: Participant dosages measured at baseline and daily until end of study (day 15), total daily dose of methadone converted to daily morphine equivalent daily dose for cancer pain and added to total daily morphine dosages. From these daily values, maximum dose recorded will be Opioid Maximum Dose (OMD). Opioid escalation index measured as described in Outcome 1 above (milligrams calculated by formula, (OMD-OSD)/days). Low index indicates achievement of adequate analgesia or appearance of uncontrollable side effects limiting upward titration over time.
Time Frame: Day 15 (+/- 3 days)
Population: No analysis possible due to small participation numbers.
Arm/Group | Morphine Only | Morphine + Methadone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event collection from baseline to end of study, 15 days (plus or minus 3 days).
Arm/Group | Morphine Only | Morphine + Methadone
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morphine Only (N=2) | Morphine + Methadone (N=2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 2 (6) | 2 (6)
DRY MOUTH (Gastrointestinal disorders) | 1 (2) | 1 (1)
EDEMA LIMBS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 2 (3) | 1 (2)
INSOMNIA (General disorders) | 1 (1) | 0 (0)
INVOLUNTARY MOVEMENT (Musculoskeletal and connective tissue disorders) | 1 (5) | 1 (4)
MEMORY LOSS (Psychiatric disorders) | 0 (0) | 1 (1)
MOOD ALTERATION (ANXIETY) (Psychiatric disorders) | 0 (0) | 1 (1)
MOOD ALTERATION (DEPRESSION) (Psychiatric disorders) | 1 (2) | 1 (4)
NAUSEA (Gastrointestinal disorders) | 2 (6) | 1 (6)
NEUROPATHY: SENSORY (Nervous system disorders) | 1 (1) | 0 (0)
NUMBNESS AND TINGLING (Nervous system disorders) | 0 (0) | 1 (1)
PAIN (General disorders) | 2 (8) | 2 (6)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 2 (6) | 1 (4)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 1 (1)
SORE MOUTH/THROAT (Gastrointestinal disorders) | 1 (3) | 1 (3)
VOMITING (Gastrointestinal disorders) | 1 (3) | 1 (4)
WATERY EYE (Eye disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study sample size is too low for any of the differences or non-differences between the groups to be statistically significant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes